CLINICAL TRIAL: NCT02923960
Title: Effect of Nutritional Products on Metabolic Parameters in Subjects With Type 2 Diabetes
Brief Title: Effect of Nutritional Products in Subjects With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: BL33
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard ONS (Active Comparator): liquid oral nutritional supplement
  Interventions: Other: Standard ONS
- Diabetes specific ONS 1 (Experimental): liquid oral nutritional supplement with novel carbohydrate blend
  Interventions: Other: Diabetes specific ONS 1
- Diabetes specific ONS 2 (Active Comparator): liquid oral nutritional supplement with novel carbohydrate blend
  Interventions: Other: Diabetes specific ONS 2

INTERVENTIONS:
Other: Standard ONS — One serving (237 ml) standard oral nutritional beverage
  Arms: Standard ONS
Other: Diabetes specific ONS 1 — One serving (237 ml) diabetes oral nutritional beverage
  Arms: Diabetes specific ONS 1
Other: Diabetes specific ONS 2 — One serving (296 ml) diabetes oral nutritional beverage
  Arms: Diabetes specific ONS 2

SUMMARY:
This is a randomized, double blinded, multi treatment, crossover study intended to compare the glycemic and insulinemic response after consuming liquid nutritional products in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subject has type 2 diabetes
* Subject is a male or a nonpregnant, nonlactating female, at least 6 weeks postpartum prior to screening visit
* Subject's BMI is > 18.5 kg/m2 and < 35 kg/m2
* If on a chronic medication such as antihypertensive, lipid lowering, thyroid medication or hormone therapy, subject has been on constant dosage for at least two months prior to screening visit
* Subject states willingness to follow protocol as described, including consumption of study product per protocol and completing any required study forms
* Participant must refrain from taking medications/dietary supplements/herbals or substances that could modulate glucose metabolism (other than oral hypoglycemic medications), or considered anabolic, or reduce weight (fat mass)

Exclusion Criteria:

* Subject is currently diagnosed with, or has a history of severe dementia or delirium, eating disorder, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures
* Subject is known to be allergic or intolerant to any ingredient found in the study products
* Subject is participating in another study that has not been approved as a concomitant study
* Subject uses exogenous insulin for glucose control, or subject states that they have been diagnosed as having Type 1 diabetes
* Subject states they have a history of diabetic ketoacidosis
* Subject is currently on a low carbohydrate or very low carbohydrate diet
* Subject states that he/she has a current infection; has had inpatient surgery, or corticosteroid treatment in the last 3 months or antibiotics in the last 3 weeks prior to screening visit
* Subject states that he/she has an active malignancy
* Subject states that he/she has had a significant cardiovascular event ≤ six months prior to screening visit; or stated history of congestive heart failure
* Subject states that he/she has end stage organ failure or is status post organ transplant
* Subject is diagnosed with chronic kidney disease, or a history of kidney issues
* Subject states they have impaired liver function, or have a history of liver disease
* Subject has an obstruction of the gastrointestinal tract precluding ingestion of the study product, inflammatory bowel disease, short bowel syndrome or other severe forms of gastrointestinal disease such as gastroesophageal reflux disease, gastroparesis, peptic ulcer disease, celiac disease, intestinal dysmotility, diverticulitis, or ischemic colitis, or any other related condition that may cause unnecessary subject discomfort
* Subject states they have a chronic, contagious, infectious disease
* Subject has taken/is currently taking any herbals, dietary supplements, or medications during the past four weeks prior to screening visit that are designed to affect blood glucose.
* Subject states that he/she has clotting or bleeding disorders
* If selected for continuous blood glucose monitoring, subject has skin lesions, hyperhidrosis, eczema, psoriasis, scarring, redness, infection or edema at the flash constant glucose monitoring application site(s) that could interfere with device placement or the accuracy of interstitial glucose measurements.
* If selected for continuous blood glucose monitoring, subject has an X-ray, MRI or CT appointment scheduled during the period of study participation, or another procedure that would require removal of the flash constant glucose monitoring sensor.
* Subjects on sulfonylureas, meglitinides, and α-glucosidase inhibitors, insulin, or subject on more than two oral hypoglycemic medications excluding aforementioned.
* Subjects on oral hypoglycemic medications that has changed in last 2 months.
* Subject's HbA1c, per point of care device is > 8%

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Plasma Glucose Concentration | 0 to 240 minutes

SECONDARY OUTCOMES:
Serum Insulin Concentration | 0 to 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Owen Kelly, PhD, Study Chair — Abbott Nutrition
Locations (2):
- United States (2):
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Radiant Research, Inc., Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Undecided